CLINICAL TRIAL: NCT03739645
Title: Physiological Studies in Healthy Subjects, Chronic Pain Patients and in Patients Undergoing Neurosurgical Procedures of Human Forebrain Mechanisms Mediating Somatic Sensation, Motor Control and Neurological Disorders
Brief Title: Human Behaviors Related to the Expectation of Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00079932; 2R56NS038493-16A1 (NIH)
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Fear Pain
Keywords: fear; pain; conditioning; skin conductance response; Ratings of Pain and Conditioning; Eye position metrics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Analysis of eye position and skin conductance levels will be examined to identify attentional and anxiety related processes for the fear of pain during the conditioned stage. Correlation of skin conductance levels versus slopes during the conditioning stage with state versus trait anxiety will be taken as confirmatory evidence. Power analysis for a two-way ANOVA was conducted to determine a sufficient sample size using an alpha of 0.05, power 0.80, a high effect size (pilot data indicate η2 values for main effects > 0.5). Based on these assumptions, we conservatively use a sample size of 40.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye position and tense arousal over time a metrics for sustained attention in conditioned fear. (Experimental): After conditioning the conditioned stimulus induces autonomic metrics like skin conductance and cognitive ratings like expectancy of the unconditioned stimulus after conditioning. Activity across blocks in the conditioning stage demonstrates that the skin conductance can produce a progressive decrease in skin conductance over the conditioning stage of our fear conditioning protocol. The decline is not apparently related to habituation or changes in the skin conducting electrodes or recording system. It does correspond to the decrease in performance of a visual fixation task which is part of the fear conditioning during the conditioning stage; and to an increase in the unpleasant psychologic activation termed tense arousal over the same stage. If both these changes are found he then we may conclude that sustained task related attention is produced during fear conditioning
  Interventions: Behavioral: Skin conductance levels and slopes over time in conditioned fear as metrics.as metrics for anxiety

INTERVENTIONS:
Behavioral: Skin conductance levels and slopes over time in conditioned fear as metrics.as metrics for anxiety — After fear conditioning the cue induces autonomic responses like skin conductance and cognitive ratings like expectancy of the unconditioned stimulus after cueing or conditioning. Activity across blocks in the conditioning stage shows that the skin conductance can be described by levels, and slopes which might be related to state anxiety and trait anxiety (Spielberger trait and state anxiety inventory or questionnaire). These skin conductance measures may be concrete metrics for psychological processes in healthy subjects. We will carry out a partial correlation analysis of levels, state anxiety and trait anxiety, and then a similar analysis of slopes, state anxiety and trait anxiety. These results may show that concrete skin conductance levels and slopes are related to metrics of subjective self report measures of state and trait anxiety.

SUMMARY:
The conditioned expectation of pain is an important aspect of pain-related disability produced by environments and stimuli associated with a painful injury on the job, although the neuroscience of this expectation is unclear. We will develop and use novel objective methods for measurement of expectation and threat related attention. The results of this study may lead to testable hypotheses regarding the psychological basis of the fear of pain, threat and task related attention. We will also use these results, and development of novel autonomic and ratings metrics for state and trait anxiety as well as threat and task related attention which could be used as an instrumented test for diagnosis and management of PTSD and anxiety disorders. .

DETAILED DESCRIPTION:
The conditioned expectation or fear of pain often results in disability produced by stimuli related to a painful injury on the job, although there are questions about attentional and anxiety related expectation. Conditioned expectation in humans can be produced by a protocol that consists of a train of two visual conditioning stimuli, one of which is paired (CS+) with a painful laser pulse unconditioned stimulus (US), while the other is not. This protocol will be used to study the expectation of pain in this study, and its relationship to task and threat related attention measured by eye position and to anxiety, task directed sustained attention, and scalp EEG metrics. These results may also be used in an instrumented test for the diagnosis and management of PTSD and anxiety disorders.

EEG studies may clarify the relationship of unpleasantness (valence) and the ability of stimuli to command attention (salience) of the conditioned and unconditioned stimuli which which are significant but under studied aspects of the fear of the pain. Studies of scalp EEG activation and functional connectivity will be used to estimate global properties of the forebrain networks involved in the fear of pain, as well as the valence and the salience) of the conditioned and unconditioned stimuli.

Activations are measured by the proportion of electrodes over a quadrant or lobe of the scalp a significant ratio of electrical power following an event over baseline (event related spectral perturbation, ERSP). Functional connectivity will be measured by causal interactions following an event over baseline. The approach of this protocol is that causal interactions are based upon causal influences by an approach based upon the concept of linear predictability. Briefly, a signal Y is said to exert an influence upon signal X when the predication error of the X is reduced by adding the past information of Y (causal interaction). The signals from any two quadrants or lobes will be analyzed by event related causality to determine the magnitude and direction of causal interactions between the two to determine fear and pain related directed interactions related to aversive conditioning.

Our Preliminary Data shows EEG activations in global distributed forebrain networks for the expectation of pain are consistent with the evidence of studies of anatomic projections and functional MRI (fMRI) signals. These models including our Preliminary Data from intracranial recordings identify structures in the medial temporal lobe (amygdala and hippocampus) which are involved in expectation of pain, while EEG suggests global activations related to valence and salience of conditioned and unconditioned stimuli. The premise of this study is that novel autonomic and eye position metrics will measure state and trait anxiety as well as threat and task related attention to parse out the experience and anticipation of pain.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 80 years of age.
* Fluent speaker of English.
* Undergoing seizure monitoring at Hopkins Hospital through intracranial electrodes.
* Possess ability to understand study procedures and comply with them for the entire length of the study;
* Women of childbearing age must use pharmacological contraception (oral or patch) for the duration of the study follow-up.

Exclusion Criteria:

* Inability or unwillingness of individual to give written informed consent. Presence of any neurological disease other than epilepsy which is unstable or is not optimally treated.
* Presence of a significant abnormality on routine neuropsychological testing.
* Presence of any medical or psychiatric disease which is unstable or is not optimally treated.

Presence of an abnormal MRI scan except for Normal variants or Medial Temporal Sclerosis (altered pathology and MRI signal in temporal lobe).

* Women who are pregnant or women of childbearing capacity who may become pregnant (i.e. not using contraception).
* Presence of generalized seizures, or reflex seizures i.e. triggered by a sensory stimulus.
* Presence of a language or hearing impairment.
* Non-English speakers.

Ages: 16 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred A Lenz, MD PhD, Principal Investigator — Dept of Neurosurgery, Hopkins University.
Locations (1):
- Hopkins Epilepsy Monitoring Unit, Zayhed 12., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI and Co-PIs are working with the Johns Hopkins Pain Research Institute to set up a website for the Institute to include the labs carrying out pain research in the Department of neurosurgery. As a part of this effort we will include the Functional Neurosurgery Lab to share the following information in the public domain: 1. Our research focus. 2. Biosketches of the investigators 3. All publications as final manuscripts at the time of acceptance for publication, 4. Funded grant applications 5. Collaborators 6. Contact information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The website will be complete in 3 years.

REFERENCES:
- [Result] Liu CC, Shi CQ, Franaszczuk PJ, Crone NE, Schretlen D, Ohara S, Lenz FA. Painful laser stimuli induce directed functional interactions within and between the human amygdala and hippocampus. Neuroscience. 2011 Mar 31;178:208-17. doi: 10.1016/j.neuroscience.2011.01.029. Epub 2011 Jan 20. PMID 21256929
- [Result] Liu CC, Chien JH, Kim JH, Chuang YF, Cheng DT, Anderson WS, Lenz FA. Cross-frequency coupling in deep brain structures upon processing the painful sensory inputs. Neuroscience. 2015 Sep 10;303:412-21. doi: 10.1016/j.neuroscience.2015.07.010. Epub 2015 Jul 10. PMID 26168707
- [Result] Chien JH, Colloca L, Korzeniewska A, Cheng JJ, Campbell CM, Hillis AE, Lenz FA. Oscillatory EEG activity induced by conditioning stimuli during fear conditioning reflects Salience and Valence of these stimuli more than Expectancy. Neuroscience. 2017 Mar 27;346:81-93. doi: 10.1016/j.neuroscience.2016.12.047. Epub 2017 Jan 8. PMID 28077278
- [Result] Liu CC, Crone NE, Franaszczuk PJ, Cheng DT, Schretlen DS, Lenz FA. Fear conditioning is associated with dynamic directed functional interactions between and within the human amygdala, hippocampus, and frontal lobe. Neuroscience. 2011 Aug 25;189:359-69. doi: 10.1016/j.neuroscience.2011.05.067. Epub 2011 Jun 12. PMID 21664438
- [Result] Liu CC, Ohara S, Franaszczuk P, Zagzoog N, Gallagher M, Lenz FA. Painful stimuli evoke potentials recorded from the medial temporal lobe in humans. Neuroscience. 2010 Feb 17;165(4):1402-11. doi: 10.1016/j.neuroscience.2009.11.026. Epub 2009 Nov 17. PMID 19925853

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 32 participants were consented. 1 participant didn't meet criteria and was not randomized.
Period: Overall Study
Arm/Group | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear.
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear.
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Skin Conductance Response
Description: Concrete metric is skin conductance response to painful laser pulse stimulus measured in microSiemens. Higher values mean more emotional arousal or stress. All participants experienced two types of conditioned stimuli, one stimulus signaled danger and the other safety. Only during the danger stimulus would the participant receive a laser pulse.
Time Frame: 5 seconds post conditioned stimulus
Measure: Mean (Standard Error); unit: micro Siemens
Arm/Group | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear.
Number analyzed (Participants) | 31
micro Siemens
  Danger Stimulus | .19 (.037)
  Safety Stimulus | .016 (.0068)

2. Primary Outcome: State Anxiety as Assessed by the Spielberger State-Trait Anxiety Inventory
Description: The Spielberger State-Trait Anxiety Inventory (STAI) is a 40-item self-report questionnaire with 20 items designed to assess State anxiety (temporary feelings of anxiety). The State anxiety score range is between 20 and 80 with higher scores representing higher anxiety. State anxiety was measured and is reported.
Time Frame: Baseline, post conditioning up to 6 minutes
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear.
Number analyzed (Participants) | 31
score on a scale
  Baseline | 36.28 (1.56)
  Post Conditioning | 39.59 (2.22)

3. Primary Outcome: Experimental Pain as Assessed by a Pain Rating Scale
Description: Pain Rating for Unpleasantness on a scale of 0 - 10 where 10 is the worst imaginable. All participants experienced two types of conditioned stimuli, one stimulus signaled danger and the other safety. Only during the danger stimulus would the participant receive a laser pulse.
Time Frame: Post conditioning approximately 6 minutes
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear.
Number analyzed (Participants) | 31
score on a scale
  Danger Stimulus | 3.43 (.59)
  Safety Stimulus | .82 (.27)

ADVERSE EVENTS:
Time Frame: Up to 3 days
Arm/Group | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear.
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eye Position and Tense Arousal Over Time a Metrics for Sustained Attention in Conditioned Fear. (N=31)
Burn (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03739645/Prot_SAP_000.pdf